CLINICAL TRIAL: NCT05691634
Title: Prospective Study Evaluating the Clinical Tolerance of Skin Tattoos During MRI Examinations (TATOU - IRM)
Acronym: TATOU - IRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Collaborators: Cimror (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A02758-33
Record Dates: First submitted 2023-01-09; First posted 2023-01-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Tattoo Disorder; MRI
Keywords: Tattoo disorder; MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with tatoo (Experimental)
  Interventions: Procedure: MRI; Other: Likert scale questionnaire

INTERVENTIONS:
Procedure: MRI — Patient with a tatoo will perform an MRI. The possible symptoms during the MRI or after MRI will then be described (duration, type,...).
Other: Likert scale questionnaire — The patient will appreciate his feeling after MRI on a Likert scale (from 1 to 5)

SUMMARY:
MRI examinations are potential sources of complications related to the displacement of ferromagnetic objects, but also to heating effects that can go as far as burns. This overheating can be caused by contact with external equipment (sensors, cables, etc.). Patients with skin tattoos may experience specific complications as tingling or "burning" felt at the site of the tattoo. They can be followed by a transient erythema with edema around the reversible tattoo in 12 and 72 hours. One observation of severe 2nd degree burns has been reported. They would be linked to the presence of metallic salts in the dermis, resulting from interactions between the pigments and the magnetic field but their mechanisms are poorly identified and divergent.

The aim of this study is to assess the rate of MRI causing complications in patients with tattoos.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* tattoo patient
* Ability to answer the questionnaire
* Affiliated patient or beneficiary of a social security scheme
* Patient having been informed and not objecting to the research

Exclusion Criteria:

* Minor
* Patient unable to understand and respond to questionnaires due to language difficulties or cognitive impairment
* Patient objecting to research
* Pregnant or breastfeeding woman
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of MRIs resulting in at least one complication in patients with tattoos. | 1 day
  Complications are defined by the occurrence of symptoms felt by the patient (tingling, stinging, burning, redness, swelling) and by the occurrence of side effects visible to the operator (redness, oedema/tumefaction, others) and confirmed by the investigator present during the examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle Santé République, Clermont-Ferrand, France